CLINICAL TRIAL: NCT01632436
Title: A Non-randomized Cohort Study With Matched Controls Investigating Pharmacokinetic Parameters and Safety of a Single Dose of Pixantrone With Metastatic Cancer and Moderate, Severe, or No Hepatic Impairment.
Brief Title: Pharmacokinetic and Safety Study of Pixantrone in Patients With Metastatic Cancer and Hepatic Impairment
Acronym: Hepatic
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No eligible patients enrolled
Sponsor: CTI BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIX 112
Record Dates: First submitted 2012-06-27; First posted 2012-07-03 (Estimated); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Metastatic Cancer
Keywords: Hepatic impairment; Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis | interventions — pixantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stage 1 -Moderate Hepatic Impairment (Experimental): Pixantrone
  Interventions: Drug: Pixantrone
- Stage 2 - Severe Hepatic Impairment (Experimental): Pixantrone
  Interventions: Drug: Pixantrone

INTERVENTIONS:
Drug: Pixantrone — Experimental Drug

SUMMARY:
This study will be conducted in patients with metastatic cancer and either moderate, severe, or no hepatic impairment who have failed other antineoplastic therapies or for whom there is no standard therapy. The study will be conducted in two stages. Using an existing pixantrone population pharmacokinetic (PPK) model, a model-based strategy will be used to evaluate the findings from the first stage of the study conducted in patients with moderate hepatic impairment and matched controls. The PPK evaluation will be completed prior to enrolling patients with severe hepatic impairment and additional matched controls during the second stage of the study. Patients with hepatic impairment will be paired with matched control patients with normal hepatic function, matched on gender, age, and body surface area (BSA).

DETAILED DESCRIPTION:
This study will be conducted in patients with metastatic cancer and either moderate, severe or no hepatic impairment who have failed other antineoplastic therapies or for whom there is no standard therapy. The study will be conducted in two stages. Stage I will include patients with moderate hepatic impairment and Stage II will include patients with severe hepatic impairment. An analysis of data from the Stage I portion of the study will be performed to decide whether to enroll patients in the Stage II portion of the study. Patients with hepatic impairment (either moderate or severe) will be paired with matched control patients with normal hepatic function, matched on gender, age, and body surface are (BSA). Patients will receive a single dose of pixantrone on day 1 of a 21 day cycle. Blood samples will be obtained at various time points during the first week of the first cycle for pharmacokinetic (PK) analysis. If any patient with hepatic impairment develops a dose limiting toxicity, subsequent patients will be administered a lower dose of pixantrone. If any patient with hepatic impairment who is receiving the reduced dose of pixantrone experiences a dose limiting toxicity, the study will be terminated. Patients who demonstrate any clinical, radiologic, or other evidence of response or stabilization after the initial dose of pixantrone and who wish to continue treatment may do so at the discretion of the Investigator. Patients receiving additional cycles will be treated with pixantrone every 21 days for up to 5 additional cycles and will be followed for safety only, until 30 days after the last dose.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Institutional Review Board (IRB) approved consent form
2. Age ≥ 18 years old
3. Histological confirmation of cancer from any previous cytological or tissue report
4. Diagnosis of metastatic disease based on biopsy, imaging, or clinical criteria
5. Failure of other antineoplastic therapies, or disease for which no standard therapy exists
6. At least 28 days since last antineoplastic therapy
7. ECOG PS ≤ 2 (see Appendix 8.2)
8. Life expectancy ≥ 12 weeks in Investigator's judgment
9. LVEF ≥ 50% by echocardiogram
10. Hemoglobin ≥ 8 g/dL (can be post transfusion)
11. Platelets ≥ 75 x 109/L
12. ANC > 1.5x109/L
13. Stage I, moderate hepatic impairment: 1.5 < total serum bilirubin ≤ 3.0 ULN Stage II, severe hepatic impairment: 3.0 < total serum bilirubin < 4.0 ULN Stages I and II, normal liver function: total bilirubin < 1.0 ULN
14. Serum creatinine ≤ 1.0 x ULN
15. All acute toxicities related to prior treatment recovered to grade ≤ 1 or baseline except alopecia
16. Willingness and ability to comply with the visit schedule and assessments required by the study protocol
17. If fertile, both males and females must agree to use appropriate and effective contraception (oral contraceptives, barrier methods, approved contraceptive implant, long-term injectable contraception, or intrauterine device) for the duration of study participation and for 6 months after last dose of study drug.

Exclusion Criteria:

1. Prior treatment with a cumulative dose of doxorubicin or equivalent exceeding 450 mg/m² according to the calculation index in Appendix 8.1
2. Total serum bilirubin > 4.0 ULN
3. LVEF < 50% by echocardiogram
4. Active grade 3/4 infection
5. Major surgery ≤ 28 days prior to first dose
6. Gilbert's syndrome
7. Known human immunodeficiency virus
8. Any antineoplastic therapy ≤ 28 days prior to first dose
9. New York Heart Association Classification III or IV heart disease (see Appendix 8.3)
10. Any contraindication or known allergy or hypersensitivity to the study drug
11. Pregnant or lactating
12. Concomitant therapy with anticancer agents (corticosteroid use is permitted)
13. Any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study procedures or follow-up schedule
14. Severe and/or uncontrolled medical disease that could compromise participation in the study or any medical or psychiatric condition that in the opinion of the Investigator would make study drug administration hazardous or obscure the interpretation of data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-05; Primary Completion 2017-08 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Cmax | Day 1 Cmax
  Cmax ratio of patients with hepatic impairment / matched control (geometric mean and 90% confidence interval)
Clearance | Day1-7
  Clearance ratio of patients with hepatic impairment / matched control (geometric mean and 90% confidence interval)
AUC | Day 1-7
  AUCss ratio of patients with hepatic impairment / matched control (geometric mean and 90% confidence interval)

SECONDARY OUTCOMES:
Incidence of Adverse Events | Day 1-7
  Safety and tolerability of pixantrone, including monitoring of adverse events (AEs); an AE is any untoward medical occurrence in a study subject administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage

CONTACTS AND LOCATIONS:
Overall Officials: John Sarantopoulos, MD, Principal Investigator — UTHSCSA- Cancer Therapy & Research Center
Locations (1):
- UTHSCSA-Cancer Therapy-Research Center, San Antonio, Texas, United States